CLINICAL TRIAL: NCT05806268
Title: Patient Characteristics, Associated Factors, and Clinical Outcomes of Prescribing Encorafenib and Binimetenib Versus Dabrafenib and Trametinib Among BRAF v600 Mutated Metastatic Melanoma Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS58
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: BRAF v600 Mutated Metastatic Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dab/tram: Patients received dabrafenib and trametinib treatment
- Enco/bini: Patients received encorafenib and binimetenib treatment

SUMMARY:
This was a retrospective real-world evidence cohort study. The study was conducted using the NOBLE (Novartis Braf+ meLanoma patients ObsErvational) dataset, with a study period from 01 January 2011 to 31 May 2020. All included patients were ≥18 years of age and were required to have a diagnosis of unresectable stage III or IV melanoma (ICD-9 172.x & ICD-10 C43 or D03x), treatment with dabrafenib and trametinib (dab/tram) or encorafenib and binimetenib (enco/bini) on or after 01 June 2018, and evidence of a BRAF-positive result prior to or up to 30 days after therapy initiation.

No quota of centers was established a priori. Given the retrospective nature of this study, all patients who met the inclusion/exclusion criteria from the NOBLE dataset were included.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of melanoma (ICD-9 172.x & ICD-10 C43 or D03x)
* Pathologic stage III (unresectable) or IV at initial diagnosis on or after 01 January 2011
* 1L treatment with enco/bini or dab/tram on or after 01 June 2018
* Evidence of a BRAF test
* Evidence of a BRAF-positive result prior to or up to 30 days after 1L therapy initiation
* At least 18 years of age at the time of initiation of 1L treatment Exclusion criteria
* Documented receipt of a clinical trial treatment for cancer at any time on or after September 2015
* Diagnosis of a second primary cancer or secondary cancer following initiation of 1L metastatic melanoma (MM) treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Assessment of clinical predictors for choice of first-line (1L) therapy between dab/tram and enco/bini | Up to approximately 2 years

SECONDARY OUTCOMES:
Percentage of patients receiving enco/bini or dab/tram in the 1L of therapy | Up to approximately 2 years
Percentage of patients switching from 1L enco/bini therapy to either another targeted therapy (TT) or second-line (2L) immunotherapy (IO) | Up to approximately 2 years
Percentage of patients switching from 1L dab/tram therapy to either another TT or IO 2L therapy | Up to approximately 2 years
Percentage of patients who discontinued treatment in 1L and associated reasons, overall and by cohort | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States